CLINICAL TRIAL: NCT03373708
Title: Prospective Randomized Controlled Study on the Risk and Clinical Benefit of Chemotherapy and Intensive Endocrine Therapy for Luminal B1 Early-stage Breast Cancer
Brief Title: Risk and Clinical Benefit of Chemotherapy and Intensive Endocrine Therapy for Luminal B1 Early-stage Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhiyong Yu (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Yu, Director of the Breast Surgery Ⅰ, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI-03
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer; Chemotherapy; Endocrine Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Epirubicin; Doxorubicin; Cyclophosphamide; Docetaxel; Goserelin; Tamoxifen; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EC follow T group (Experimental): Epirubicin 100mg/m2 on day 1 cyclophosphamide 600mg/m2 on day1 every 2 weeks for four cycles followed by docetaxel 100mg/m2 on day 1 every 3 weeks for four cycles
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- TC follow endocrine (Experimental): Docetaxel 75mg/m2 on day 1 and cyclophosphamide 600mg/m2 on day 1 every 3 weeks for four cycles followed by goserelin acetate+tamoxifen for young patients/ letrozole for postmenopausal patients
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Goserelin acetate; Drug: Tamoxifen; Drug: Letrozole

INTERVENTIONS:
Drug: Epirubicin — 100mg/m2
  Other Names: Adriacin
  Arms: EC follow T group
Drug: Cyclophosphamide — 600mg/m2
  Other Names: Cyclophosphamide injection
Drug: Docetaxel — 75mg/m2(TC), 100mg/m2(EC-T)
  Other Names: Docetaxel injection
Drug: Goserelin acetate — 3.6mg every month
  Other Names: Zoladex
  Arms: TC follow endocrine
Drug: Tamoxifen — 10mg twice daily oral
  Other Names: Nolvadex
  Arms: TC follow endocrine
Drug: Letrozole — 2.5mg every daily oral
  Other Names: Femara
  Arms: TC follow endocrine

SUMMARY:
Breast cancer is the most common female malignancy in the world, and the leading cause of cancer-associated mortalities among women. Hormone receptors (HR) including ER and PR are the main prognostic factor for breast cancer patients. Breast cancer subtype was defined by ER, PR, HER2 and Ki67 status since the definition of intrinsic subtypes for breast cancer. Breast cancer which ER are positive have less aggressive and better long-term prognoses than other breast cancer subtype. Luminal B1 was definited as ER Positive, PR positive <20%, or Ki-67 ≥20% , and HER2-Negative. Although standard therapy to HR positive breast cancer is endocrine treatment, evidence reported that Luminal B1 breast cancers with lower PR expression are less sensitive to tamoxifen than luminal A breast cancers with higher PR expression, and the specific mechanism is not clear. We previously had a clinically analysed, and we found the Luminal B1 breast cancer had a significant proportion with 38%. Whether we need standard chemotherapy or chemotherapy based intensive endocrine therapy for those patients? In our research, we divided the patients with ER positive, PR negative, and HER-2 negative into two groups. One groups will be treated with 8 cycles of chemotherapy (EC×4-T×4). The other received 4 cycles of chemotherapy (TC×4) then will be given the intensive endocrine therapy (Goserelin acetate+Tamoxifen for young patients/Letrozole for postmenopausal patients). The primary endpoint is to assess disease-free survival (DFS) and overall survival (OS) in different regiments, the secondary endpoint is to assess the expression of female hormone levels. The correlation of the expression of female hormone levels with the clinical outcomes, so that the investigators could optimize adjuvant treatment regiment with luminal B1 breast cancer.

DETAILED DESCRIPTION:
The trial is designed to investigative the risk and clinical benefit of chemotherapy and intensive endocrine therapy for Luminal B1 early-staged breast cancer. In this trial the investigators will randomly assign 200 primary breast cancer patients to receive four cycles of epirubicin and cyclophosphamide (EC) followed by four cycles of docetaxel(T), or four cycles of docetaxel and cyclophosphamide (TC) followed by intensive endocrine therapy (Goserelin acetate+Tamoxifen/Letrozole for young patients) . Patients with HER-2 positive was excluded. The patient's conditions will be assessed before, and after every four cycles of adjuvant chemotherapy to determine if there is any progression of the disease. The patient's conditions will be assessed every three months when they received the intensive endocrine therapy (Goserelin acetate+Tamoxifen for young patients/Letrozole for postmenopausal patients). Patients will be followed up for DFS and OS in different regiments, the secondary endpoint is to assess the expression of female hormone levels. The correlation of the expression of female hormone levels with the clinical outcomes, so that the investigators could optimize adjuvant treatment regiment with luminal B1 breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* All patients were required to give written informed consent.
* Patients present with operable breast cancers that were diagnosed by histopathology and have no distant metastasis.
* Have no history of anti-cancer therapies including chemotherapy, radiation therapy, hormone therapy and surgical therapy
* Have normal cardiac functions by echocardiography
* ECOG scores are ≤ 0-1.
* Patients are disposed to practice contraception during the whole trial.
* The results of patients' blood tests are as follows:

Hb ≥ 90 g/L WBC ≥ 3.0×109/L Plt ≥ 100×109/L Neutrophils ≥ 1.5×109/L ALT and AST ≤ 2.5 times of normal upper limit. TBIL ≤ 1.5 times of normal upper limit. Creatinine ≤ 1.5 times of normal upper limit.

* ER+ Her2- early-stage breast cancer

Exclusion Criteria:

* Have other cancers at the same time or have the history of other cancers in recent five years, excluding the controlled skin basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of cervix.
* Active infections
* Severe non-cancerous diseases.
* The patients are undergoing current administration of anti-cancer therapies, or are attending some other clinical trails.
* Inflammatory breast cancer.
* Pregnant or lactational, or patients refuse to practice contraception during the whole trial.- Page 5 of 5 -
* The patients are in some special conditions that they can't understand the written informed consent, such as they are demented or hawkish.
* Have allergic history of the chemotherapeutic agents.
* Bilateral breast cancers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2017-12-20 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  To determine the percentage of disease-free survival (DFS) for the EC follow T arm and TC follow endocrine therapy arm separately.

SECONDARY OUTCOMES:
Expression of female hormone levels | 5 years
  To assess the association between the female hormone levels and the clinical outcomes
Overall survival (OS) | 5 years
  To determine the percentage of Overall survival (OS) for the EC follow T arm and TC follow endocrine therapy arm separately.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Yu, PhD, Study Chair — Shandong Cancer Hospital and Institute; Zhaoyun Liu, MD, Principal Investigator — Shandong Cancer Hospital and Institute